CLINICAL TRIAL: NCT05788952
Title: UNRAVEL - The Role of Intestinal and Vaginal Microbiota, Estrogenic Activity, Metabolic Profile & Nutritional Status in Symptom Severity and Quality of Life of Portuguese Women With Endometriosis - an Exploratory Study
Brief Title: The Role of Intestinal and Vaginal Microbiota, Estrogenic Activity, Metabolic Profile & Nutritional Status in Endometriosis
Acronym: UNRAVEL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Academia CUF (Unknown)
Responsible Party: Sponsor
Other Study IDs: UNRAVEL
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Endometriosis
Keywords: Endometriosis; Gut microbiota; Vaginal microbiota; Estrogenic activity; Xenoestrogens; Metabolic biomarkers; Nutritional status
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometriosis (EMs) is one of the most prevalent benign gynaecological diseases, and it is an inflammatory oestrogen-dependent condition. Several authors have proposed that anatomical, genetic, endocrine, immunological, environmental, hormonal, and inflammatory factors may influence tissue implantation outside the uterus. An approach to EMs aetiology that involves defining a profile to the vaginal and gut microbiota, estrogenic activity, and exposure to xenoestrogens and also metabolic and nutritional status of women with EMs may help identify some important patterns to better characterize this disease and also to define more personalized nutritional strategies, also predicting patients' predisposition to therapy success. This is an observational study on premenopausal woman, diagnosed with EMs, who will be recruited on the outpatient gynaecology appointment, to evaluate the vaginal and intestinal microbiome, measure the total estrogenic activity, assess the metabolic biomarkers and the nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Premenopause;
* Diagnose of endometriosis by clinical and/or imaging criteria (associated adenomyosis is accepted);
* BMI between 18.5 and 30.0 kg/m2

Exclusion Criteria:

* Postmenopause;
* Vegetarian diet;
* Pregnancy or breastfeeding;
* Continuous hormonal therapy for endometriosis;
* Laparoscopic surgery for endometriosis purpose;
* Gastrointestinal or vaginal infections;
* Intaken antibiotics and/or probiotics within the last 8 weeks;
* Medications to treat vaginal infections in the past 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any premenopausal woman diagnosed with endometriosis under an outpatient gynaecology appointment at one of the recruitment locations.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal microbiome | day 1
  Characterization of the vaginal microbiome. Bacterial DNA will be extracted from cytology samples. 16S rRNA gene will be sequenced by next-generation sequencing (NGS). All the identified bacterial phyla, genus and species will be expressed in percentage.
Intestinal microbiome | day 1
  Characterization of the intestinal microbiome at baseline. Bacterial DNA will be extracted from fecal samples. 16S rRNA gene will be sequenced by next-generation sequencing (NGS). All the identified bacterial phyla, genus and species will be expressed in percentage.
Strogen levels | day 1
  Mean/median of total and free estrone (E1) and estradiol (E2) (ng E2-equivalents L-1) at baseline.
Fasting blood glucose | day 1
  Mean/median of fasting blood glucose levels (mg/dL) levels at baseline.
Insulin | day 1
  Mean/median of insulin (μU/mL) levels at baseline.
Total cholesterol | day 1
  Mean/median of total cholesterol (mg/dL) levels at baseline.
HDL cholesterol | day 1
  Mean/median of high-density lipoprotein (HDL) cholesterol (mg/dL) levels at baseline.
LDL cholesterol | day 1
  Mean/median of low-density lipoprotein (LDL) cholesterol (mg/dL) levels at baseline.
25-hydroxy vitamin D | day 1
  Mean/median of 25-hydroxy vitamin D (ng/mL) levels at baseline.
Ascorbic acid | day 1
  Mean/median of ascorbic acid (umol/L) levels at baseline.
Alpha (α)-tocopherol | day 1
  Mean/median of α-tocopherol (ug/mL) levels at baseline.
Omega-3 index | day 1
  Mean/median of omega-3 index (uL) levels at baseline.

SECONDARY OUTCOMES:
Quality of life questionnaire | day 1
  Median of quality of life by the Quality of Life Scale (QOLS) questionnaire at baseline. The QOLS is a 16-item questionnaire and consists of 7 different subscales. The total score is calculated as the sum of the 16 items each ranged from 0 to 7. The final score ranges from 16 to 112 points (lower scores indicate more unfavourable conditions).
Symptoms severity | day 1
  Median of symptoms severity by the Numerical Rating Scale (NRS) at baseline. The NRS is a scale that assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Diana Teixeira, PhD, Principal Investigator — NOVA Medical School | Faculdade de Ciências Médicas, Universidade Nova de Lisboa
Locations (1):
- NOVA Medical School|Faculdade de Ciências Médicas, Universidade NOVA de Lisboa, Lisbon, Portugal